CLINICAL TRIAL: NCT02666625
Title: Study of Iatrogenic Effects of Treatment for Childhood Cancer - Constitution of a Biological Samples Bank as Part of a Cohort of Patients (Cohort FCCSS)
Brief Title: Iatrogenic Effects of Treatment for Childhood Cancer Constitution of a Biological Samples Bank
Acronym: BIO-F
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-A00555-34; 2010/1623 (Other: CSET number)
Record Dates: First submitted 2015-08-03; First posted 2016-01-28 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Paediatric Malignancies
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated for cancer in childhood
  Interventions: Procedure: saliva samples; Procedure: blood samples

INTERVENTIONS:
Procedure: saliva samples
Procedure: blood samples

SUMMARY:
The constitution of a biological samples bank, attached to epidemiological studies Cohort F-CCSS on iatrogenic effects of treatment of childhood cancer, will identify genetic variants that can modulate the iatrogenic risks of these treatments. The main objective is to provide a biological samples bank to consider, besides the carcinogenic risks, the risk of other iatrogenic diseases in these children, in particular cardiac, cerebrovascular, lung, bone and kidney. These conditions can be very incapacitating and in some cases, fatal. Their impact, however, is poorly estimated as occurring in adulthood, they are rarely made in relation to the treatment received in childhood. The overall project is expected to eventually better define the iatrogenic effects prevention strategies for cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for a first cancer in childhood
* Adult patients
* Signed informed consent
* Patient insured or enjoying a social security scheme

Exclusion Criteria:

* Minor patients
* Under legal protection measure patients
* Refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for a paediatric malignancies before the year 2000 having survived two years after treatment of solid tumor diagnosed before 18 years old
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2010-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Study of genetic factors who might lead to secondary iatrogenic pathology due to treatment of a childhood cancer | seven years

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne, France